CLINICAL TRIAL: NCT00365326
Title: Safety and Efficacy of Autologous, Intracoronary Stem Cell Injections in Total Coronary Artery Occlusions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Collaborators: University Hospitals Cleveland Medical Center (Other); Arteriocyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HFM-705
Record Dates: First submitted 2006-08-15; First posted 2006-08-17 (Estimated); Last update posted 2022-03-24 (Actual); Status verified 2006-08

CONDITIONS: Coronary Occlusion
Keywords: AC133; coronary; bone marrow; autologous; coronary artery disease
MeSH Terms: conditions — Coronary Occlusion; Coronary Artery Disease

ARMS (1):
- Treatment with autologous bone marrow (BM)-derived CD133+ stem cell therapy (Experimental): The Phase I single arm clinical study, was designed to assess the safety and feasibility of a dose escalating intracoronary infusion of autologous bone marrow (BM)-derived CD133+ stem cell therapy to the patients with chronic total occlusion (CTO) and ischemia.
  Interventions: Biological: Catheter-based intracoronary injection

INTERVENTIONS:
Biological: Catheter-based intracoronary injection — This Phase I single arm clinical study, was designed to assess the safety and feasibility of a dose escalating intracoronary infusion of autologous bone marrow (BM)-derived CD133+ stem cell therapy to the patients with chronic total occlusion (CTO) and ischemia. Nine patients were received CD133+ cells into epicardial vessels supplying collateral flow to areas of viable ischemic myocardium in the distribution of the CTO.

SUMMARY:
This phase I clinical trial will evaluate the safety and efficacy of intra-coronary injection of AC133 selected autologous marrow-derived stem cells in patients with chronic coronary artery occlusion. A clinical study to determine the therapeutic potential of marrow-derived stem cells as an adjunct therapy to current standard therapies for CAD is warranted. The current initiative is to investigate a model of chronic myocardial ischemia and (1) to determine whether intra-coronary injection of selected autologous marrow-derived AC133 stem cells is reasonably safe for use in humans and (2) if this treatment shows any improvement in coronary perfusion, as assessed using non-invasive imaging. This study is structured to evaluate the feasibility and safety of autologous AC133+ bone marrow-derived stem cell via intra-coronary injection into documented ischemic but viable myocardial zones via established collateral vessels. The epicardial vessel that normally supplies the ischemic zone must be 100% chronically occluded and considered non-revascularizable by percutaneous means.

DETAILED DESCRIPTION:
This study is composed of one phase. The objective of Phase I is to assess the safety and feasibility of performing escalating doses of autologous AC133+ selected bone marrow-derived stem cell with intracoronary infusion via epicardial vessels supplying collateral flow to areas of viable ischemic myocardium in the distribution of a chronic totally occluded vessel. Additionally, focus on the assessment of the benefit achieved from the infusion of stem cells and subsequent angiogenesis at 6 months will be observed.

Potential candidates are patients with a known total occlusion of an epicardial vessel, with a documented chronically ischemic territory supplied by collateral conduits.

Secondary Objectives include:

1. Improvement in ETT as determined by: total exercise duration on the 6 month ETT in seconds time to: onset of angina, one mm ST depression, onset of angina or one mm ST depression (whichever occurs first)
2. Reduction in the area of ischemia will be evaluated by nuclear (sestamibi) stress imaging with exercise or pharmacologic stress.
3. Improvement in viability within the chronically ischemic zone as measured by nuclear (sestamibi) stress imaging.
4. Improvement in angina as per Angina Questionnaire (The Seattle Angina Questionnaire) at 7, 14, 30, 90, 180, and 365 days.
5. Major adverse cardiac events (MACE) assessment (composite endpoint including cardiac death, myocardial infarction, ischemia-driven target vessel revascularization, CABG, CVA, and rehospitalization for angina), MACE definitions:

   Myocardial Infarction (All ST segment elevation MIs as diagnosed on electrocardiogram by a staff cardiologist and all non-ST segment elevation MIs as defined by elevation in cardiac enzyme markers per the hospital laboratory guidelines) Cerebral Vascular Accidents (e.g., acute neurological event).
6. Concomitant Medication usage (e.g., changes in utilization of PRN or sublingual nitroglycerin for angina)
7. ECG changes at day of discharge, 7, 14, 30, 90, 180, and 365 days.
8. Functional capacity (e.g., exercise duration (time) and changes in METS achieved on treadmill study at 6 month follow-up).
9. Echocardiogram assessment of left ventricular ejection fraction and regional wall motion abnormalities at 180 days (e.g., changes in regional wall motion score and/or changes in left ventricular ejection fraction).

ELIGIBILITY:
Inclusion Criteria:

1. The patient must have at least one region of chronically ischemic myocardium formerly perfused by a coronary artery which is now 100% occluded and not revascularizable by conventional percutaneous or surgical methods.
2. Well-established collateral vessels at least 1.5-mm luminal diameter by coronary angiography to the chronically ischemic myocardium must be identified at the time of diagnostic coronary angiography.
3. Evidence of viable myocardium in the area supplied by collateral conduits intended for stem cell infusion must be demonstrated by nuclear (sestamibi) stress imaging.
4. Left ventricular ejection fraction of >45% as per 2D echocardiogram.
5. Patient must experience class II - IV angina as defined by the Canadian Cardiovascular Society (CCS).
6. Patient will be followed by the investigating team over the 12 month follow-up period.
7. The patient must be at least 18 years of age and have signed an informed consent.
8. If the patient is a female of child-bearing potential, a pregnancy test is negative.

Exclusion Criteria:

Patients meeting any of the following exclusion criteria will be excluded from the study:

1. Patient with coronary lesions amenable to percutaneous coronary intervention including brachytherapy, or where CABG is indicated.
2. Any contraindication for cardiac catheterization and percutaneous coronary intervention as per institutional guidelines.
3. Any contraindication for bone marrow aspiration as per institutional guidelines.
4. Myocardial infarction within the previous 3 months.
5. Documented bleeding diathesis.
6. Known malignancy involving the hematopoietic/lymphoid system.
7. Patients with baseline ECG abnormalities that would hinder interpretation of baseline ECG uninterpretable for ischemia (e.g., left bundle branch block, left ventricular hypertrophy with strain pattern, Wolff-Parkinson-White syndrome).
8. Patients with severe co-morbidities including renal failure (serum creatinine > 2.0).
9. Anticipated unavailability for follow-up visits secondary to psychological or social reasons.
10. NYHA class III or IV congestive heart failure
11. Anemia with hemoglobin concentration < 8 mg/dl
12. Thrombocytopenia with platelet count < 100 x 103

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2006-01; Primary Completion 2007-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Assess the safety and feasibility of performing autologous AC133+ selected bone marrow-derived stem cell intra-coronary infusion and determine whether any benefit is achieved from the infusion of stem cells by non-invasive cardiac assessment. | 7days-6months
  Determine whether intra-coronary injection of selected autologous marrow-derived AC133 stem cells is reasonably safe for use in humans

SECONDARY OUTCOMES:
Improvement in ETT, reduction in ischemic area, viability improvement (nuclear stress imaging), improvement in angina (Seattle Angina Questionnaire), major adverse cardiac events assessment, echocardiogram assessment of left %EF and regional wall motion. | 7 days-6months
  Determine if this treatment shows any improvement in coronary perfusion, as assessed using non-invasive imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Dale Adler, MD, Principal Investigator — Case Western Reserve University; Hillard Lazarus, MD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States